CLINICAL TRIAL: NCT02676050
Title: Exploratory Study to Optically Visualise Activated Neutrophils and the Proto-oncogene, c-MET, in Lung Cancer Using DUAL Colour Fibre-based Endomicroscopy
Brief Title: Visualising c-MET and Activated Neutrophils in Lung Cancer
Acronym: DUAL
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: C-met marker expired
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DUAL
Record Dates: First submitted 2016-02-02; First posted 2016-02-08 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging agents and imaging devices (Experimental): All participants in Cohort 1 will be dosed on one occasion with the optical imaging agents and Cohort 2 can be dosed twice per agent. The final dosage will be <100ug per agent. The agents will be delivered using a novel delivery catheter and imaged with a novel imaging fibre and microendoscopy system.
  Interventions: Other: Optical Imaging Agents (EMI-137, NAP); Device: Delivery Device Cathetar and Miniaturised imaging fibre; Device: Optical endomicroscopy system

INTERVENTIONS:
Other: Optical Imaging Agents (EMI-137, NAP) — Both optical imaging agents (NAP and EMI-137) will be administered to each patient during a bronchoscopy procedure. A novel delivery catheter (to deliver both agents), imaging fibre and endomicroscopy system with viewer software will be used to detect c-MET and activated neutrophil signal in the human lung.
  Other Names: EMI-137, NAP
Device: Delivery Device Cathetar and Miniaturised imaging fibre — Both optical imaging agents (NAP and EMI-137) will be administered and imaged simultaneously during a bronchoscopy procedure using the devices mentioned above.
Device: Optical endomicroscopy system — The signal emitted by both optical imaging agents (NAP and EMI-137) will be visualised using a novel endomicroscopy system.

SUMMARY:
Lung cancer is currently a major health problem in the UK. Despite being one of the most common cancers, lung cancer has a poor prognosis compared to other types of cancer and is the leading cause of cancer death in the world. As opposed to other organs, the lung is highly susceptible to inflammatory insults, for example from bacterial infection-induced and tobacco-induced inflammation. It has long been known that the cellular microenvironment that nurtures tumour growth and development is linked to sites of chronic inflammation but molecular insights into how external inflammation boosts or inhibits cancer in the lungs remains unclear. This study aims to directly visualise the expression of a well known marker of cancerous tissue, c-MET, and the activity of neutrophils in human lung cancer in vivo in situ using fibre-based endomicroscopy.

DETAILED DESCRIPTION:
The primary objective of this study is to directly deliver a microdose of two optical imaging agents to 20 patients with suspected or confirmed lung cancer to assess whether the agents can detect c-MET expression and neutrophil activity in human lung cancer.

The primary endpoint is to visualise the delivery of these imaging agents to assess imaging parameters in patients with suspected or diagnosed lung cancer using a novel delivery catheter, imaging fibre and fibre-based endomicroscopy system.

This protocol will involve two cohorts of patients; Cohort 1 will include patients scheduled for resection of their lung cancer and Cohort 2 will be patients with suspected inoperable stage 3/4 lung cancer scheduled for a diagnostic bronchoscopy followed by therapy. For both cohorts, eligibility will be verified by a clinical trial physician after written informed consent has been obtained.

Fibre-based endomicroscopy (FE) will be performed and up to 100μg of both optical imaging agents will be instilled during a bronchoscopy procedure. CT identified regions of architecturally normal lung in all participants will act as internal controls and will be used to compare the signal in normal and diseased lung tissue. Tissue samples taken from both cohorts will be collected for ex vivo validation including immunohistochemistry, zymography and genomic screening.

A cardiorespiratory exam, chest x ray and routine observations will be performed 4-6 hours following the administration of both imaging agents. All participants will be visited by a member of the research team 24 hours (± 4 hours) after dosing to ensure no adverse events were experienced. All participants in Cohort 1 will complete the study when the 24 hour assessment has been successfully completed and all adverse events have been resolved. Participants in Cohort 2 will be invited back for a second bronchoscopy following the first round of their therapy to investigate whether the expression of c-MET or the level of neutrophil activity has changed. All participants in Cohort 2 will complete the study when the second 24 hour assessment has been successfully completed and all adverse events have been resolved.

ELIGIBILITY:
INCLUSION CRITERIA FOR COHORT 1 • Patients undergoing cardiothoracic surgery for resection of lung cancer

INCLUSION CRITERIA FOR COHORT 2

• Patients with inoperable stage 3 or 4 lung cancer

INCLUSION CRITERIA FOR BOTH COHORTS

* ≥ 16 years
* Provision of informed consent from the patient prior to any study related procedures.
* Normal electrocardiogram (ECG)
* Forced Expiratory Volume (FEV1) >1L
* Thoracic CT scan taken in the last 20 weeks
* Attending consultant permission for bronchoscopy
* Readily accessible target areas with bronchoscopy and FE

EXCLUSION CRITERIA

* Refusal for participation by attending consultant
* Unsuitable for bronchoscopy
* Any history of anaphylaxis
* Significant coagulopathy, which causes bronchoscopy to be unsuitable, as determined by clinical co-investigator or the participant's attending consultant, using information which is routinely available
* Myocardial infarction in the preceding four weeks
* Women who are pregnant or are breastfeeding
* Receiving drugs that cause increased autofluorescence in the lung, specifically amiodorane and methotrexate
* Oxygen saturation <92% breathing room air
* Platelet count < 50 x 109/L
* Bleeding diathesis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
The measurement of optical agents in the lung | On average, fluorescence signal can be detected within 5 minutes following optical imaging agent administration.
  The primary endpoint of this clinical investigation is to image the delivery of the optical imaging agents in human lung cancer using a novel delivery catheter, imaging fibre and fibre-based endomicroscopy system.

SECONDARY OUTCOMES:
Quantification of signal of imaging agents | On average, fluorescence signal can be detected within 5 minutes following optical imaging agent administration.
  To determine whether neutrophil activation and c-MET activity are increased in human lung cancer in vivo in situ
Ability of novel device to deliver agents and image simultaneously | Within 5 minutes
  To determine if the novel delivery catheter can co-deliver imaging agents and image simultaneously
Whether expression correlates with treatment response | Within 4-6 weeks following first round of therapy
  To establish if neutrophil activity and c-MET upregulation can predict stage 3/4 tumour response to either chemotherapy or radiotherapy (Cohort 2).

CONTACTS AND LOCATIONS:
Overall Officials: Kev Dhaliwal, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No